CLINICAL TRIAL: NCT06392373
Title: Skeletal Muscle Recovery From Aerobic Exercise During Acute High Altitude Exposure When Consuming Carbohydrate Compared to Carbohydrate Plus Protein
Brief Title: High Altitude Muscle Recovery
Acronym: HAMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-04H
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: High Altitude
MeSH Terms: conditions — Altitude Sickness | interventions — CVS 1123

STUDY DESIGN:
Intervention Model Description: Double blinded randomized crossover design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate plus protein (Experimental): Study beverages consumed over the initial 3 hours recovery phase from aerobic exercise, consuming 0.9g CHO/kg/hr + 0.3g PRO/kg/hr during high altitude exposure.
  Interventions: Dietary Supplement: CHO+PRO
- Carbohydrate (Active Comparator): Study beverages consumed over the initial 3 hours recovery phase from aerobic exercise, consuming1.2g CHO/kg/hr during high altitude exposure.
  Interventions: Dietary Supplement: CHO

INTERVENTIONS:
Dietary Supplement: CHO+PRO — 0.9 g CHO/kg/hr + 0.3 g PRO/kg/hr
  Arms: Carbohydrate plus protein
Dietary Supplement: CHO — 1.2 g CHO/kg/hr
  Arms: Carbohydrate

SUMMARY:
To understand alterations in glycogen and molecular regulation of skeletal muscle glucose uptake, glycogen synthesis, and muscle protein recovery when consuming CHO (glucose) or CHO+PRO (glucose + whey) post-exercise during unacclimatized high altitude exposure, randomized crossover double blinded studies will be conducted in the hypobaric/hypoxic chamber at USARIEM Table 1. Briefly, the study consists of a 2 day baseline period at SL followed by two, 3 day trial periods (with the 3rd day being a testing day) at HA. The baseline is separated from trial 1 for a least a day, and trial 1 & 2 separated by at least 4 days. Volunteers will consume CHO (glucose) or CHO+PRO (glucose + whey) drinks post-exercise during unacclimatized high altitude exposure during the two trial periods. The order of the drinks will be randomized (using a random number generator such as randomizer.org) and kept by a study staff not directly involved in data collection to maintain blinding.

DETAILED DESCRIPTION:
Dietary strategies that restore muscle glycogen and promote muscle repair and remodeling in recovery from exercise are needed to protect muscle mass and sustain performance during strenuous military operations conducted at high altitude (HA; > 2500 m elevation). However, most military personnel who operate at HA are native lowlanders and, thus, unacclimatized to the hypoxemia that occurs upon initial HA exposure. We demonstrated that acute HA exposure (within 5 hours) dysregulates peripheral glucose uptake and inhibits post-exercise muscle anabolism in lowlanders sojourning at 4,300 m. Our results suggest that traditional recommendations to consume solely carbohydrate immediately post-exercise to facilitate muscle recovery may be inadequate for lowlanders exercising within the first several hours of HA exposure. In a recent meta-analysis by our group, we reported that the effects of ingesting carbohydrate (CHO) compared to isocaloric carbohydrate plus protein (CHO+PRO) on muscle glycogen repletion were equivocal, yet the combined macronutrient blend confers an additional metabolic advantage than CHO alone because it stimulates muscle repair/remodeling by upregulating anabolic signaling and protein synthesis. Our findings suggest post-exercise CHO intake can be reduced in place of an isocaloric amount of PRO when exercising at HA without comprising glycogen repletion. However, whether CHO+PRO promotes post-exercise glycogen repletion and muscle anabolism as compared to CHO alone when peripheral glucose uptake and anabolic signaling are dysregulated with acute HA exposure has not been determined. This study aims to determine the effects of ingesting CHO or an isocaloric amount of CHO+PRO post-aerobic exercise on glycogen synthesis, molecular regulation of glucose uptake, storage, and muscle protein synthesis during acute HA exposure. This study will employ a randomized crossover double-blinded design and be conducted in the hypobaric/hypoxic chamber at USARIEM. A total of 10 healthy, physically active men and women between the ages of 18-39 years will be studied. Following 48 hours of controlled exercise and diet to normalize muscle glycogen stores, volunteers will report to the laboratory after a 10-h overnight fast. After a muscle biopsy is taken from the vastus lateralis at baseline, volunteers will be brought to HA (460 mmHg) conditions within the hypobaric/hypoxic chamber at USARIEM and complete a standardized glycogen depletion protocol on a cycle ergometer. After completing the glycogen depletion exercise a second muscle biopsy will be taken. Volunteers will then consume 1.2 g CHO/kg/h or 0.9 g CHO/kg/h + 0.3 g PRO/kg/h over a 3-h recovery period. A third and fourth biopsy will be taken 4 and 6 hours into recovery to characterize the molecular regulation of glucose uptake, glycogen synthesis, and muscle protein synthesis over time. Serial blood draws will be collected during each trial to assess endocrine and circulating substrate responses in CHO and CHO+PRO. Trials will be separated by a minimum of 4 days. The primary risks associated with this study include those associated with acute hypobaric hypoxia, exercise, muscle biopsies, and blood draws.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 - 39 years
* Physically active (exercise minimum 2-4 days per week)
* Have supervisor approval (permanent party military and civilians at NSSC)
* Willing to refrain from alcohol, nicotine products and dietary supplement use during the study
* Females must have normal menstrual cycles between 26-32 days in duration; 5 menstrual cycles within the past 6 months; or using oral/hormonal contraceptive use which contains low-dose estrogen/progesterone to maintain continuous levels throughout the 28-day cycle (i.e., no placebos)
* Only consume caffeine products during the study if provided by study staff

Exclusion Criteria:

* Born at altitudes greater than 2,100 m (Subjects will inform the study team if they were born in Eagar AZ, Mammoth Lakes CA, CO, NM, UT, or WY).
* Musculoskeletal injuries that compromise exercise capability
* Metabolic or cardiovascular abnormalities, or gastrointestinal disorders (e.g. hypothyroidism, cardiovascular disease, Crohn's disease, etc.)
* Taking medication that affects macronutrient metabolism and/or the ability to participate in strenuous exercise (e.g. thyroxine, beta blockers, insulin etc.)
* Living in areas that are more than 1,200 m, or traveled to areas that are more than 1,200 m for five days or more within 2 months of data collection (e.g. Idaho Falls, ID; Denver, CO; etc.)
* Prior diagnosis of high-altitude pulmonary edema or high-altitude cerebral edema
* Presence of asthma or respiratory tract infections
* Smoking or vaping (other forms of nicotine users, i.e., chewing tobacco will not be excluded; individuals who quit smoking or vaping for more than 90 days may be included)
* Taking medications that interfere with oxygen delivery and transport (e.g. albuterol, EPO, etc.)
* Hematocrit (HCT) <41% and Hemoglobin (HBG) <13.5 g/dL(Males), HCT <36% and HBG <12.0 g/dL (Females), and Sickle Cell Anemia/Trait
* Whole blood donation within 8 weeks of the study
* Unwilling or unable to only consume study diets or foods provided due to personal preference, dietary restrictions, and/or food allergies
* Unwilling or unable to adhere to study physical restrictions (abstain from exercise or recreational activities i.e., pick-up basketball during the study procedures)
* Pregnant, trying to become pregnant, and/or breastfeeding (results of urine pregnancy test or self-report for breastfeeding will be obtained before body composition testing)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Muscle Glycogen Concentrations | 6 hours
  Determine the effects of of consuming a CHO (1.2 g CHO/kg/hr) compared to an isocaloric CHO+PRO (0.9 g CHO/kg/hr + 0.3 g PRO/kg/hr) supplement on post exercise muscle glycogen concentrations (umol/kg dry muscle weight) during the initial 6 hours of aerobic exercise recovery
Phosphorylation status of rpS6 | 6 hours
  Determine the effects of of consuming a CHO (1.2 g CHO/kg/hr) compared to an isocaloric CHO+PRO (0.9 g CHO/kg/hr + 0.3 g PRO/kg/hr) supplement on post exercise muscle the fold change in the phosphorylation of rpS6 during the initial 6 hours of aerobic exercise recovery

CONTACTS AND LOCATIONS:
Locations (1):
- USARIEM, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT06392373/ICF_000.pdf